CLINICAL TRIAL: NCT06865222
Title: Variable Pulse Transcranial Magnetic Stimulation for Treatment of Post COVID Syndrome
Brief Title: Post COVID-19 Syndrome Treatment With Variable Pulse Transcranial Magnetic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ryan T. Hurt, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-011546
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Post COVID-19 Condition
MeSH Terms: interventions — estramustine-binding protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anosmia (Experimental): Subjects Olfactory Threshold Test scores correspond to Anosmia or Hyposmia
  Interventions: Procedure: Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) - 2 weeks
- Tinnitus (Experimental): Subjects have >0 score on Tinnitus Handicap Inventory (not present prior to COVID infection)
  Interventions: Procedure: Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) - 2 weeks
- Fatigue (Experimental): Subjects have Total Modified Fatigue Impact Scale (MFIS) Score of 40 or above
  Interventions: Procedure: Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) - 4 weeks

INTERVENTIONS:
Procedure: Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) - 2 weeks — The Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) will be administered through an FDA-approved Transcranial Magnetic Stimulation (TMS) medical device. Results of the baseline EEG will be uploaded to NoetherTech's EMBP software on the Mayo Clinic campus, and transferred to Noethertech servers for TMS parameter determination
  TMS treatment will be one 30 min session per day, 5 days per week (Monday-Friday), for 2 weeks.
  Arms: Anosmia; Tinnitus
Procedure: Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) - 4 weeks — The Electromagnetic Brain Pulsing Variable Pulse Protocol (EMBP) will be administered through an FDA-approved Transcranial Magnetic Stimulation (TMS) medical device. Results of the baseline EEG will be uploaded to NoetherTech's EMBP software on the Mayo Clinic campus, and transferred to Noethertech servers for TMS parameter determination
  TMS treatment will be one 30 min session per day, 5 days per week (Monday-Friday), for 4 weeks.
  Arms: Fatigue

SUMMARY:
The purpose of this study is to test if Variable Pulse TMS (Transcranial Magnetic Stimulation) can result in objective improvements in patients with Post COVID Syndrome (PCS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a recent episode of COVID-19 and who present to the Post COVID-19 Clinic at Mayo Clinic Rochester with at least one of the PCC symptoms of interest - anosmia, tinnitus, fatigue. Symptoms consistent with PCC lasting at least 1 month after the positive test date. Subjects must have ongoing symptoms for > 4 weeks following the start of an acute covid infection. This is consistent with the CDC definition for post covid conditions. Start date is determined by date of first positive COVID test. There is no limitation of maximum time from acute infection start.
* At least one of the PCC symptoms of interest:

  * Anosmia: Olfactory Threshold Test scores corresponding to Anosmia or Hyposmia
  * Tinnitus: >0 score on Tinnitus Handicap Inventory (not present prior to SARS-COVID 2 infection)
  * Fatigue: Total Modified Fatigue Impact Scale (MFIS) Score of 40 or above

Exclusion Criteria:

* Implanted electronic devices, including pacemakers, defibrillators, implant medication pumps, or vagus nerve stimulators (VNS)
* Active alcohol abuse: >14 drinks a week or formal diagnosis, illicit drug use or drug abuse
* Any seizure history within the past 10 years
* Intracranial implant within 30 cm of magnet (e.g., aneurysm clips, endovascular coil, cerebral shunts, brain stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed
* Enrolled or plans to enroll in an interventional trial during this study
* Previous stroke with residual deficits
* Subjects unable to comprehend or follow verbal commands
* Subjects unable to comprehend and sign the informed consent
* Based on PI's or local physician's assessment that subject unable to tolerate the trial procedure due to medical condition
* Clinical abnormality or clinically unstable medical condition, as indicated by medical history, physical examination, or clinical laboratory testing, that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results
* Pregnant or trying to become pregnant; negative urine pregnancy test at screening will be required for females of childbearing potential
* Any condition which in the judgment of the investigator would prevent the subject from completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in University of Pennsylvania Smell Identification Test (UPSIT) Olfactory Threshold Test score | Baseline, 2 weeks, 10 weeks
  Subjects in the Anosmia group will be assessed using the the University of Pennsylvania Smell Identification Test (UPSIT) test is commercially available booklet of 40 scratch-and-sniff odors, arranged in microencapsulated "scratch and sniff" format. Each correct identification is worth one point, with a score of 40 indicating a perfect smell. It has been used for the assessment of anosmia in COVID-19.
Change in Tinnitus Handicap Inventory Scale score | Baseline, 2 weeks, 10 weeks
  Subjects in the Tinnitus group will be assessed using the Tinnitus Handicap Scale (THI) is a 25-item questionnaire that assesses the severity of tinnitus. The THI is scored using a 5-point Likert Scale. The THI total score ranges from 0 to 100, with a higher score indicating a greater handicap from tinnitus.
Change in Modified Fatigue Impact Scale score | Baseline, 4 weeks, 12 weeks
  Subjects in the Fatigue group will be assessed using the Modified Fatigue Impact Scale (MFIS) is scored using a 5-point Likert scale. The scale ranges from 0 to 4, with 0 = 'Never' to 4 = 'Almost always'. The total obtainable score is 20. Higher scores indicate greater fatigue.

SECONDARY OUTCOMES:
Change in General Anxiety Disorder-7 (GAD-7) score | Baseline, 12 weeks
  The General Anxiety Disorder 7-item (GAD 7) scale will assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety.
Change in Patient Health Questionnaire-9 score | Baseline, 12 weeks
  The Patient Health Questionnaire 9-item (PHQ-9) scale used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.
Change in PROMIS Global-10 score | Baseline, 12 weeks
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Change in alpha wave characteristics measured via EEG. | 1 week, 12 weeks
Number of serious adverse events (SAEs) | 2 years
  Number of occurrences of serious adverse events (SAEs) throughout the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T. Hurt, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No